CLINICAL TRIAL: NCT05156606
Title: T&T Trial: Adding Testosterone to Tamoxifen in Male Breast Cancer Patients
Brief Title: Testosterone & Tamoxifen Trial
Acronym: T&T
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Five patients were included; it did not succeed in recruiting the target number of 6 patients. This is as a result of the rarity of this disease in men.
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100318
Record Dates: First submitted 2021-11-16; First posted 2021-12-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Male Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male | interventions — Testosterone

STUDY DESIGN:
Intervention Model Description: Male patients with metastatic BC (n=6)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): After the baseline imaging with FES- and FDHT-PET is completed, tamoxifen 20mg 1dd1 (standard dosage) plus testosterone (Androgel®) will be started. The first 3 patients will receive 25mg testosterone once daily (half the standard starting dosage for male hypogonadism). If this is well tolerated after 3 weeks, the dosage will be increased to 50mg once daily. Out of precaution, the safety profile of the 50mg dosage in the first 3 patients will be evaluated after all 3 patients have received 50mg testosterone for 2 cycli (8 weeks), prior to proceeding to the next 3 patients. Patients will be treated with tamoxifen and testosterone until disease progression or unacceptable toxicity.
  Interventions: Drug: AndroGel

INTERVENTIONS:
Drug: AndroGel — After the baseline imaging with FES- and FDHT-PET is completed, tamoxifen 20mg 1dd1 (standard dosage) plus testosterone (Androgel®) will be started. The first 3 patients will receive 25mg testosterone once daily (half the standard starting dosage for male hypogonadism). If this is well tolerated after 3 weeks, the dosage will be increased to 50mg once daily. Out of precaution, the safety profile of the 50mg dosage in the first 3 patients will be evaluated after all 3 patients have received 50mg testosterone for 2 cycli (8 weeks), prior to proceeding to the next 3 patients. Patients will be treated with tamoxifen and testosterone until disease progression or unacceptable toxicity.

SUMMARY:
This is a concise single arm, feasibility study, which will be executed in the University Medical Center Groningen, The Netherlands. Male patients with metastatic BC (n=6) are eligible for this study after at least 1 line of conventional endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. A history of proven ER+ (>10% of cells), AR+ (>10% of cells), and HER2- metastatic BC
3. Tumor progression after at least one line of conventional endocrine therapy (tamoxifen, AI, fulvestrant, CDK4/6, ±LHRH analogue).
4. Age ≥ 18 years
5. Adequate hematological, renal and liver function as follows:

   * Absolute neutrophil count > 1.5 x 109/L
   * Platelet count >100 x 109/L
   * White blood cell count >3 x 109/L
   * AST and ALT <2.5 or <5.0 in case of liver metastases x upper limit of normal (ULN)
   * Creatinine clearance >50mL/min
   * Prothrombin time, partial thromboplastin time and INR <1.5 x ULN
6. Written informed consent

Exclusion Criteria:

1. History of prostate, testicular or liver cancer
2. Patients already using testosterone supplements
3. Patients using medication with anti-androgenic effects (e.g. spironolactone)
4. Elevated PSA (>4μg/L) or severe urinary tract problems (as defined with a Prostate Symptom Score >19). Patients with known BRCA mutation and PSA >3 μg/L will be referred to the urologist for prostate cancer screening, and can participate if they have no signs of prostate cancer.
5. Hematocrit >50%
6. Patients with uncontrolled hypertension, diabetes mellitus or other significant cardiovascular morbidity.
7. Patients with recent history of coronary artery disease or trombo-embolic events within 6 months prior to screening
8. Severe concurrent disease, infection, co morbid condition that, in the judgment of the investigator would make the patient inappropriate for enrollment
9. Visceral crisis and/or rapid progression necessitating chemotherapy
10. Previous allergic reaction to androgen agonists
11. Contra-indication for PET imaging
12. Tamoxifen or fulvestrant treatment <5 weeks prior to FES-PET.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male breast cancer patients
Enrollment: 5 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Safety profile | At 8 weeks and follow-up through study completion, an average of 1 year
  Safety profile, defined as the number of AEs and SAEs that occur while on tamoxifen and testosterone treatment.

SECONDARY OUTCOMES:
AR to ER ratio | At baseline
  AR to ER ratio on baseline FES- and FDHT-PET imaging (assessed per lesion and per patient by quantitative analysis using standardized uptake values (SUV)) and/or tumor tissue (assessed by percentage of ER and AR expression).
Treatment response | 8 weeks
  Treatment response on 8 weeks FDG-PET/CT (assessed per lesion and per patient by quantitative analysis using standardized uptake values (SUV).
Imaging and response | At 8 weeks and follow-up through study completion, an average of 1 year
  Relation between baseline imaging and tumor characteristics to treatment response.
Adverse events based on dosages | At 8 weeks and follow-up through study completion, an average of 1 year
  Difference in adverse events between the two testosterone dosages.

CONTACTS AND LOCATIONS:
Overall Officials: Geke A.P. Hospers, MD,PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands